CLINICAL TRIAL: NCT06533319
Title: Screening and Treatment for Chronic Hepatitis C Infection of Persons Incarcerated in the County Jail Setting
Brief Title: Hepatitis C Treatment in Idaho County Jails
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Idaho Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-US-342-7112
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Intervention Model Description: Multi-site, prospective cohort study at Idaho county jails with quantitative methods and survey.
Masking Description: All study components will be blind to individuals in charge of the study, with the exception of the prescribing clinician and primary investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients infected with chronic hepatitis C who are also incarcerated in an Idaho county jail (Other): Patients infected with chronic hepatitis C who are also incarcerated will be enrolled into the study and provided FDA approved Epclusa (sofosbuvir/velpatasvir) for treatment of chronic hepatitis C. Epclusa (sofosbuvir/velpatasvir) is currently used as a first line treatment for chronic hepatitis C. This study will focus on effectiveness of treatment in the county jai setting.
  Interventions: Drug: sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir — Patients who qualify for the study will be provided with sofosbuvir/velpatasvir for chronic hepatitis C treatment.

SUMMARY:
To explore the feasibility of opt in Hepatitis C Virus (HCV) screening and initiation of HCV treatment during incarceration in county jails including;

1. incarcerated persons positive for HCV who remain in jail for duration of 12 weeks of treatment and
2. incarcerated persons positive for HCV in jails less than the duration of 12 weeks of treatment who receive remaining supply of study drug on discharge with appropriate linkage to care.

Assess quality of life measures in participants being treated for their HCV through the validated questionnaire EuroQol-5D at baseline and post-treatment.

DETAILED DESCRIPTION:
Aligning with the World Health Organization (WHO) global guidance and recommendation to eliminate viral hepatitis by 2030 will require designated focus on priority populations who are disproportionately impacted by viral hepatitis. Addressing chronic hepatitis C virus (HCV) with the justice involved population is crucial in reducing HCV within the greater population. Inmate populations bear a disproportionate share of the burden of HCV infection. HCV prevalence is 10-20 fold greater in the incarcerated population than the general population, although wider uptake among people who are incarcerated remains limited. Addressing HCV in the incarcerated population is a strategy to bring the US closer to successfully eradicating the HCV epidemic. Additionally, previous qualitative research has suggested that justice involved individuals felt incarceration is an apt time to initiate treatment and is a missed opportunity to not do so, and that waiting and initiating treatment upon release faces multiple challenges, including insurance or Medicaid enrollment, making appointments, transportation and work commitments.

HCV in the jail setting is a public health issue that needs to be addressed. Extensive modelling has shown that HCV testing in people who are incarcerated prevents community spread of HCV and is cost effective. Furthermore, there is guidance and recommendations for HCV testing in the prison system where a vast majority of research is being conducted. However, there is limited guidance for HCV testing within jails. Thus, county jails are critical partners, and potentially may serve as an important setting for HCV screening, diagnosis and treatment, although data is scarce in this realm. We therefore aim to explore whether county jails are a practical and feasible setting for HCV screening, and initiating HCV treatment, including whether an incarcerated person resides in the county jail for the duration of treatment (group 1), or is released to the community in the midst of treatment with a supply of remaining study drug and linked to appropriate care (group 2).

ELIGIBILITY:
Inclusion Criteria:

* All participants greater than 18 years old and incarcerated in an Idaho county jail greater than 10 days.
* All participants who are not sentenced to prison terms at Idaho Department of Corrections (IDOC). Participants sentenced to IDOC will receive screening and treatment per IDOC policy.
* Participants diagnosed with HCV and qualify for the AASLD Simplified Treatment Algorithm for Treatment Nave Adults Without Cirrhosis.

Exclusion Criteria:

* All participants greater than 18 years old and incarcerated in an Idaho county jail greater than 10 days.
* All participants who are not sentenced to prison terms at Idaho Department of Corrections (IDOC). Participants sentenced to IDOC will receive screening and treatment per IDOC policy.
* Participants diagnosed with HCV and qualify for the AASLD Simplified Treatment Algorithm for Treatment Nave Adults Without Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response | 12 weeks after treatment
  Undetectable hepatitis C RNA

SECONDARY OUTCOMES:
Quality of life improvement | At study enrollment and 12 weeks after treatment
  Improvement in quality of life measures after treatment of hepatitis C as measured by SF-12 tool